CLINICAL TRIAL: NCT01100749
Title: Demography, Clinical Characteristics, Metabolic Status, Viral Subtype and Genetics of Infection With Hepatitis C Genotype 3 in Canada
Brief Title: Chronic Hepatitis C (CHC) - Genotype 3 Infection in Canada
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Geno3-Demographics Study
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Hepatitis C - Genotype 3
Keywords: Hepatitis C; Genotype 3; Demographics; Genetics; Metabolic status
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples will be collected for DNA extraction. Also, blood specimens will be collected for genotype subtype analysis and HOMA score calculation.
Oversight: Data Monitoring Committee: No

SUMMARY:
Hepatitis C is a small RNA virus spread by blood to blood contamination. There are to date 6 known genotypes and within each there are several subtypes. Although all genotypes are distributed worldwide some are more common in certain countries and/or among certain populations.

DETAILED DESCRIPTION:
Genotype 3(G3) infection is the predominant type in South East Asia (Bangladesh, Pakistan, India and Sri Lanka). In addition, because of the "promiscuous exposure" to hepatitis C amongst injection drug users, it is not unusual for the latter to be infected with G3 as well. There are several subtypes of G3. Viral genotype has long been recognized as a major factor influencing the response to interferon-based therapy. Patients infected with G2 and G3 respond much better to current therapy with peginterferon and ribavirin than those infected with G1 and G4. Most studies have grouped patients with G2 and G3 together, with few published comparisons of rates of viral clearance between these two favourable genotypes.

More recently it has become evident that in all individuals with chronic hepatitis C, the presence of insulin resistance, with or without the accompanying metabolic syndrome, is a major factor which influencing the response to antiviral therapy in CHC.

Very recently it has been reported and confirmed by several sites worldwide that specific polymorphisms of the IL28 gene are closely correlated with response to antiviral therapy in genotype 1 CHC. Interestingly, the polymorphisms were also shown to segregate according to ethnicity and may explain, at least in part, the marked differences in treatment response between different ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Infected with only genotype 3, hepatitis C
* Treatment naïve before current course of therapy
* Age 18 or older

Exclusion Criteria:

* Under age 18
* Co-infection with HIV or Hepatitis B or any other HCV genotype in addition to genotype 3
* Prior treatment for Hepatitis C aside from herbal remedies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects across Canada with chronic hepatitis C, genotype 3 infection who are treatment naïve.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Factors associated with treatment outcome in genotype 3 in CHC | Within 12 weeks before starting treatment compared to end of treatment response
  To study how factors such as viral subtype, ethnicity, insulin resistance, IL28 genotype and severity of liver disease contribute to treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. E.J. Heathcote, MD, FRCP, FRCP(C), Principal Investigator — University Health Network - Toronto Western Hospital
Locations (2):
- Canada (2):
  - Toronto General Hospital - Dr. M. Sherman Liver Clinic, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Freshwater DA, O'Donnell K, Mutimer DJ. Inferior response of Asian vs non-Asian hepatitis C genotype 3 infection to combination antiviral therapy. J Viral Hepat. 2008 Feb;15(2):115-9. doi: 10.1111/j.1365-2893.2007.00899.x. PMID 18184194
- [Background] Isharwal S, Misra A, Wasir JS, Nigam P. Diet & insulin resistance: a review & Asian Indian perspective. Indian J Med Res. 2009 May;129(5):485-99. PMID 19675375